CLINICAL TRIAL: NCT02832505
Title: Applications of MRI in Kidney Disease
Status: Withdrawn | Type: Observational
Why Stopped: due to the risk for the patient and later funding issues
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1603M85321
Record Dates: First submitted 2016-06-15; First posted 2016-07-14 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease; End-stage Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-CKD (Control): Patients without CKD (eGFR ≥ 60 ml/min/1.73 mm2) (non-CKD controls).
  No intervention but only observational.
  Interventions: Other: No intervention but only observational
- CKD (chronic kidney disease): Patients with Patients with moderate to severe CKD (eGFR ranging from 26 to 44 ml/min/1.73 mm2).
  No intervention but only observational.
  Interventions: Other: No intervention but only observational
- ESRD (end-stage renal disease): Patients with advanced CKD (eGFR < 15 ml/min/1.73 mm2), preparing for or undergoing the standard thrice-weekly HD or standard PD treatment (end-stage renal disease (ESRD) patients).
  No intervention but only observational.
  Interventions: Other: No intervention but only observational

INTERVENTIONS:
Other: No intervention but only observational — This study is a cross-sectional and observational MRI study with three cohorts of patients, and no interventions will be applied.

SUMMARY:
This study has two major purposes:

1. To test developed multiple anatomic and functional MRI methods;
2. To evaluate the potentials of these MRI methods in the diagnosis, prognosis, and monitoring of the progression of renal dysfunction.

These purposes will be achieved by performing pilot studies with cohorts of patients.

DETAILED DESCRIPTION:
This study is observational with no intervention applied for the patients. In this study, multiple anatomic and functional MRI methods will be performed with three cohorts of patients. In addition to anatomic MRI methods, non-contrast enhanced functional MRI methods will also be applied to evaluate tissue perfusion and vascular reactivity in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking as primary language
2. Able to complete an approximately 75 to 90 minute cognitive and/or physical tests
3. Capable to consent to studies

Exclusion Criteria:

1. Acute psychiatric illness that would impede cognitive testing
2. Active chemical dependence, such as alcohol, narcotics or other drugs
3. Legally blind or unable to complete cognitive tests due to visual loss or deafness
4. Renal transplant recipient at time of screening or baseline
5. Severe CI unable to complete the Modified Mini-Mental State Examination [3MSE]
6. Chronic and acute pulmonary disease

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include three main cohorts of patients: 20 ESRD patients with their transition to dialysis treatment, 20 CKD controls and 20 non-CKD controls. Based on the investigators previous experience, about 20% of recruited subjects may not be able to finish the proposed studies. Therefore, a conservative estimate of the total number of subjects to be recruited is 72.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
MRI measured perfusion for each patient group | Baseline
  MRI measurements will be summarized for each patient group by using mean and standard deviation or standard error.

CONTACTS AND LOCATIONS:
Overall Officials: Xiufeng Li, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No